CLINICAL TRIAL: NCT06994481
Title: Comparison of the Effects of Endotracheal Intubation and Laryngeal Mask Applications on Optic Nerve Diameter in Pediatric Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Marmara University Pendik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, dilara gocmen, dilara göçmen, Marmara University Pendik Training and Research Hospital
Other Study IDs: marmaraeah1
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Optic Nerve Sheath Diameter; Pediatric Anesthesia; Intubation; Laryngeal Mask Airways
Keywords: optic nerve sheath diameter; pediatric patients; intubation; laryngeal mask airway

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- intubated patients: Patients aged 1-11 years who are scheduled for elective surgery and undergo endotracheal intubation
  Interventions: Diagnostic Test: optic nerve sheet diameter measurement
- group laryngeal mask airway: Patients aged 1-11 years who are scheduled for elective surgery and who use supraglottic airway devices
  Interventions: Diagnostic Test: optic nerve sheet diameter measurement

INTERVENTIONS:
Diagnostic Test: optic nerve sheet diameter measurement — Both groups will undergo bilateral optic nerve sheath diameter measurement with ultrasonography after induction, after airway manipulations, and before awakening.

SUMMARY:
This clinical study aims to investigate the effects of breathing tubes, which we use to connect children aged 1-11 to a respiratory device under general anesthesia in the operating room, on intracranial pressure after they are inserted. No changes will be made to routine anesthesia practices for this purpose, and eye examinations will be performed with an USG device. This study has no undesirable effects or risks. This study does not include any invasive procedures. You have the right to refuse to participate in the study. You have the right to withdraw from the study at any time. If you decide not to participate in the study for any reason, there will be no disruption to your treatment. You will not be liable for any financial loss if you participate in the study, and you will not be paid. Your identity will be kept confidential if you participate in the study.

DETAILED DESCRIPTION:
Our study will be conducted in the Marmara University Basibüyük Additional Service Building Prof. Dr. Asaf Ataseven Hospital Operating Room, on 200 ASA 1-2 (American Society of Anesthesiologists) children aged 1-11 who will undergo elective surgery under general anesthesia, with informed consent forms obtained from their families.

The patients will be divided into 2 groups, 100 each aged 1-4 and 4-11, and each group will be divided into two groups again, with half of them receiving an LMA (Laryngeal mask = supraglottic upper airway device) and the other half receiving an ETT (endotracheal tube).

The demographic data (age, gender, height, weight) of the patients included in the study will be recorded in the study form.

Pediatric patients included in the study will undergo standard ASA monitoring (ECG, spO2, noninvasive blood pressure, etCO2). After general anesthesia induction, intubation or LMA will be applied according to the anesthesiologist's decision. Anesthesia will be maintained with sevoflurane and remifentanyl infusion at 2% concentration in a mixture of 40% 02 and 60% air, and the inhaled sevoflurane concentration will be targeted to maintain the BIS score between 40 and 60. Peak inspiratory pressure will be kept between 11 and 13 cm H2O in order not to affect ICP.

After covering the eyes of each patient with a sterile film sheet, a thick layer of water-soluble ultrasound transmission gel will be applied to the upper eyelid, then the probe will be gently placed on the eyelid without applying pressure.

For sonographic measurements, a linear 6-13 Hz probe (Fujifilm Sonosite, Bothwell, USA) will be used at three different time points. The probe will be carefully moved to find the best image of the optic nerve entering the globe, and ONSD (optic nerve sheath diameter) will be measured 3 mm posterior to the globe. These measurements will be taken at 3 times: (TO) immediately after anesthesia induction, (T1) within a few minutes after endotracheal intubation / LMA insertion, and (T2) immediately after extubation.

At the specified times, ultrasonographic measurements will be made and recorded by 2 different individuals who have received USG training and who have previously measured the optic nerve sheath diameter. Mean arterial pressure and EtCO2 values will also be recorded simultaneously.

ELIGIBILITY:
Inclusion Criteria:

1. Classified as American Society of Anesthesiologists (ASA) physical status I or II,
2. Aged between 1 and 11 years,
3. Scheduled to receive general anesthesia,
4. Planned to be ventilated via endotracheal intubation or laryngeal mask airway (LMA).

Exclusion Criteria:

1. Families who do not provide informed consent,
2. Patients with a tracheostomy,
3. History of previous intracranial surgery (e.g., tumor resection or shunt placement),
4. History of preoperative seizures,
5. Presence of craniofacial deformities that may prevent accurate optic nerve sheath diameter (ONSD) measurement,
6. Infection, wound, or any other condition in the measurement area that may interfere with ONSD assessment,
7. Presence of conditions that may increase intracranial pressure and affect ONSD measurement (e.g., tumor, encephalitis, meningitis, or intracranial infection),
8. Patients who require a change in the endotracheal tube or laryngeal mask airway (LMA) size during the operation, or who undergo a second intubation or insertion attempt,
9. Patients who withdraw from the study.

Ages: 1 Year to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: ASA I-II children aged 1-11 years who are planned to receive general anesthesia, intubation or LMA insertion will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
optic nerve sheet diameter measurement | (TO) immediately after anesthesia induction, (T1) within a few minutes after endotracheal intubation / LMA insertion, (T2) immediately after extubation.
  For sonographic measurements, a linear 6-13 Hz probe (Fujifilm Sonosite, Bothwell, USA) will be used at three different time points. The probe will be carefully moved to find the best image of the optic nerve entering the globe, and ONSD (optic nerve sheath diameter) will be measured 3 mm posterior to the globe. These measurements will be taken at 3 times: (TO) immediately after anesthesia induction, (T1) within a few minutes after endotracheal intubation / LMA insertion, and (T2) immediately after extubation.
  At the specified times, ultrasonographic measurements will be made and recorded by 2 different individuals who have received USG training and who have previously measured the optic nerve sheath diameter. Mean arterial pressure and EtCO2 values will also be recorded simultaneously.

CONTACTS AND LOCATIONS:
Overall Officials: tümay umuroglu, professor doctor, Study Director — Marmara University

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol